CLINICAL TRIAL: NCT06934070
Title: The Predictive Value of the Albumin-Bilirubin Score and the C-Reactive Protein-Albumin-Lymphocyte Index for the Prognosis of Patients With Hepatocellular Carcinoma After Radical Resection
Brief Title: Predictive Value of Albumin - Bilirubin Score and CRP - Albumin - Lymphocyte Index for HCC Prognosis After Radical Resection
Status: Active, not recruiting | Type: Observational
Sponsor: Qiang Xu (Other)
Responsible Party: Sponsor-Investigator, Qiang Xu, Jiangxi Provincial Cancer Hospital, Jiangxi Provincial Cancer Hospital
Organization: Jiangxi Provincial Cancer Hospital (Other)
Other Study IDs: 2025ky158
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC); Hepatocellular Carcinoma (HCC) Prognosis
Keywords: HCC; Hepatocellular Carcinoma; Albumin-Bilirubin Score; CALLY; ALBI; Hepatocellular carcinoma (HCC) prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluate the predictive value of the CALLY index and ALBI grading for the prognosis of patients with hepatocellular carcinoma (HCC) after radical resection, so as to provide a reference for clinical treatment.

DETAILED DESCRIPTION:
China bears a heavy burden of liver cancer. In 2022, there were 370,000 new cases and 320,000 deaths, ranking 4th in incidence and 2nd in mortality among malignant tumors. HCC, accounting for over 80% of primary liver cancer, also has high incidence and fatality rates. Radical resection, the main cure method, has a 5-year recurrence rate over 60%, so identifying recurrence risk factors is crucial. Previously, the Child - Pugh score was used for liver function evaluation, but its assessment of ascites and hepatic encephalopathy was subjective. Quantitative systems like MELD also had limitations. Over 80% of HCC develops from cirrhosis, and inflammatory and immunonutritional indices are important in cancer development. NLR, PLR, etc., show inconsistent predictive power, and the CALLY index, though better, needs improvement. Bilirubin is a key predictor, and ALBI grading can precisely quantify liver function, related to HCC recurrence and survival. This study combines ALBI and CALLY to create a four - dimensional system, expected to reflect HCC recurrence risk. As this combined prediction research is scarce, this study evaluates their predictive value for HCC patients after radical resection, guiding clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old (2) Postoperative pathological examination confirmed hepatocellular carcinoma (HCC) (3) No other anti-tumor treatment was received before surgery (4) Radical resection was performed, and the pathological examination under the microscope showed negative surgical margins.

Exclusion Criteria:

* (1) Complicated with other malignant tumors. (2) Incomplete clinicopathological data and prognostic information. (3) Received preoperative anti-cancer treatment. (4) Follow-up less than 1 month after hepatectomy. (5) Patients with surgical contraindications before surgery, such as portal vein tumor thrombus and distant metastasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma (HCC) patients who underwent radical resection of hepatocellular carcinoma and sought medical treatment at Jiangxi Provincial Cancer Hospital
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-16 (Estimated)

PRIMARY OUTCOMES:
Recurrence - free survival period | Patients who underwent hepatocellular carcinoma resection from Jan 2018 to Jan 2025 were recruited. The time from resection to tumor recurrence or end of follow - up was measured, with calculation cutoff in Apr 2025 and a maximum of 88 months.
  It is the time interval from the patient's surgical resection to tumor recurrence or the end of follow - up. Early recurrence is defined as a tumor - free survival time of less than 2 years.

SECONDARY OUTCOMES:
Overall Survival | Patients who underwent hepatocellular carcinoma resection from Jan 2018 to Jan 2025 were collected. Survival calculation was cutoff in Apr 2025. Measurement started from the initial radical resection until death, up to 88 months.
  The length of time from either the start of treatment or diagnosis until the death of the patient from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China